CLINICAL TRIAL: NCT05161611
Title: The Effect of Oral Zinc Sulfate on Jaundice in Neonates Admitted to Neonatal Intensive Care Unit: A Randomized, Double-Blind, Clinical Trial
Brief Title: Effect of Oral Zinc Sulfate on Jaundice in Neonates Admitted to Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mariam Rajab, Chairperson of Pediatrics Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 22062021
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Serum Bilirubin
MeSH Terms: interventions — Zinc Sulfate; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc sulfate (Experimental): Patients will receive 10mg/day zinc sulfate along with phototherapy after being diagnosed to have hyperbilirubinemia
  Interventions: Drug: Zinc sulfate; Other: Phototherapy
- Placebo (Placebo Comparator): Patients will receive placebo in addition to phototherapy
  Interventions: Other: Placebo; Other: Phototherapy

INTERVENTIONS:
Drug: Zinc sulfate — 10 mg of oral zinc sulfate will be given to neonates per day
  Arms: Zinc sulfate
Other: Placebo — 10 mg of normal saline will be given to neonates per day
  Arms: Placebo
Other: Phototherapy — Neonates will be put under phototherapy

SUMMARY:
A randomized double-blind clinical trial will be performed in the neonatal intensive care unit of Makassed General Hospital in Beirut, Lebanon from December 2021 till August 2022. Randomized opaque envelopes to allocate the treatment will be used. The study will include neonates aged between 26 and 42 gestational weeks, who require phototherapy in the neonatal intensive care unit. Patients will be randomized into two groups.Both groups will receive standard conventional phototherapy, but the intervention group will receive 10 mg per day oral zinc sulfate until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Infants (post-menstrual age ≥ 26 weeks) delivered by Cesarean section or vaginal delivery.
* Diagnosed to have hyperbilirubinemia:

Hyperbilirubinemia is defined as:

* for term and near-term neonates (neonates less than 35 weeks' gestation): Serum Total Bilirubin (STB) level that would qualify for phototherapy requirement as described in American Academy of Pediatrics 2004's guidelines or absolute STB level L 15 mg/dL;
* for preterm neonates (< 35 weeks' gestation): STB level > 1% of body weight

Exclusion Criteria:

* Infants less than 26 weeks postmenstrual age
* Allergy to zinc sulfate
* Any reaction seen after administration of first dose of zinc sulfate.
* Any contraindication to oral medication
* Infants with a history of taking phenobarbital by their mother

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Phototherapy duration | Within one week
  The number of days the neonates required phototherapy

SECONDARY OUTCOMES:
Total serum bilirubin level | Within one week
  Level of total serum bilirubin will be measured in neonates
Occurrence of side effects | Within one week
  The incidence of side effects such as vomiting, diarrhea, or rash will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Rajab, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon